CLINICAL TRIAL: NCT01652599
Title: Eltrombopag and High-dose Dexamethasone as First Line Treatment for Immune Thrombocytopenia
Brief Title: Eltrombopag and High-dose Dexamethasone as First Line Treatment for IT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, David Gomez Almaguer, MD, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HE12-010
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Eltrombopag; Dexamethasone; High-dose; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eltrombopag and dexamethasone (Experimental)
  Interventions: Drug: Eltrombopag and dexamethasone

INTERVENTIONS:
Drug: Eltrombopag and dexamethasone — Eltrombopag 50 mg PO days 5-32 Dexamethasone 40 mg PO days 1-4
  Other Names: Revolade

SUMMARY:
The purpose of this study is to determine the response rate and response duration with the combination of eltrombopag and high-dose dexamethasone

DETAILED DESCRIPTION:
Immune Thrombocytopenia is an autoimmune disorder characterized by formation of autoantibodies against platelet antigens leading platelet destruction.

Corticosteroids increase the platelet count in about 80 percent of patients.However, many patients have a relapse when the dose of corticosteroid is reduced. Debilitating side effects are common in patients who require long-term corticosteroid therapy to maintain the platelet count. Eltrombopag, it is a small molecule agonist of the c-mpl (TpoR) receptor, which is the physiological target of the hormone thrombopoietin, has been shown to be effectively raise the platelet count in adult patients (aged 18 years and over) who have had their spleen removed or where splenectomy is not an option and have received prior treatment with corticosteroids or immunoglobulins, and these medicines did not work (refractary ITP). There are a few case reports where eltrombopag was an option as first line treatment for IT.

The purpose of this study is to determine the response rate and response duration with the combination of eltrombopag (50mg PO once a day for 4 weeks) and high-dose dexamethasone (40mg PO days 1,2,3,4) in untreated adult patients immune thrombocytopenic or in patients with less than 7 days of treatment with corticosteroids.

A complete platelet response is defined as an increase in platelet counts to >150×109/L on two consecutive occasions. A partial response is defined as an increase in the platelet count to between 50 and 150×109/L on two consecutive occasions, 1 week apart. Duration of response is considered from the day of the initial administration to the first time of relapse (platelet count <30×109/L)or to time of analysis.

At the end of the first 5 weeks, the patients will followed by 6 months every month.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed immune thrombocytopenic (IT) Platelet count less than 30,000/mm3 on two occasions. Platelets >30000/mm3 with bleeding.
* Less than seven days taking corticosteroids
* Normal to increased numbers of megakaryocytes on bone marrow examination in patients ≥ 60 years
* Subject is ≥ 18 years
* Subject has signed and dated written informed consent.
* No sepsis or fever
* No active infection requiring therapy
* No active chronic viral infection
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

Exclusion Criteria:

* Performance status above or equal to 2.
* Previous treatment with eltrombopag
* Immunosuppressive treatment within the last month
* Previous splenectomy
* Presence of malignant haematological disease
* Connective tissue disease
* Autoimmune hemolytic anemia
* Pregnancy and lactation
* Not willing to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with sustained response after 6 months | 6 months
  Number of patients with complete response at month 6

SECONDARY OUTCOMES:
Number of patients with complete response at month 6 | month 6
  Number of patients with platelet count at least 150x109/L, 6 months after therapy
Bleeding | month 6
  Number of patients with bleeding complication therapy

CONTACTS AND LOCATIONS:
Overall Officials: David Gomez-Almaguer, MD, Principal Investigator — Hospital Universitario Dr. Jose E. Gonzalez
Locations (1):
- Hospital Universitario "Dr. Jose E. Gonzalez" UANL, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Bussel JB, Provan D, Shamsi T, Cheng G, Psaila B, Kovaleva L, Salama A, Jenkins JM, Roychowdhury D, Mayer B, Stone N, Arning M. Effect of eltrombopag on platelet counts and bleeding during treatment of chronic idiopathic thrombocytopenic purpura: a randomised, double-blind, placebo-controlled trial. Lancet. 2009 Feb 21;373(9664):641-8. doi: 10.1016/S0140-6736(09)60402-5. PMID 19231632
- [Background] Jenkins JM, Williams D, Deng Y, Uhl J, Kitchen V, Collins D, Erickson-Miller CL. Phase 1 clinical study of eltrombopag, an oral, nonpeptide thrombopoietin receptor agonist. Blood. 2007 Jun 1;109(11):4739-41. doi: 10.1182/blood-2006-11-057968. Epub 2007 Feb 27. PMID 17327409
- [Derived] Gomez-Almaguer D, Herrera-Rojas MA, Jaime-Perez JC, Gomez-De Leon A, Cantu-Rodriguez OG, Gutierrez-Aguirre CH, Tarin-Arzaga L, Hernandez-Reyes J, Ruiz-Arguelles GJ. Eltrombopag and high-dose dexamethasone as frontline treatment of newly diagnosed immune thrombocytopenia in adults. Blood. 2014 Jun 19;123(25):3906-8. doi: 10.1182/blood-2014-01-549360. Epub 2014 May 6. PMID 24802773